CLINICAL TRIAL: NCT01194661
Title: Neural Dynamics and Connectivity in Response Inhibition and Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency); National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100185; 10-N-0185
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2017-11-16

CONDITIONS: Traumatic Brain Injury; Stroke; Headache; PTSD
Keywords: Inhibitory Control; Executive Function; fMRI; TMS; TBI; Traumatic Brain Injury; Healthy Volunteer; HV
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Headache; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Background:

- Previous research has shown that certain parts of the brain are involved in voluntarily stopping an ongoing motor response (movement); however, it is not known whether this same network is also involved in suppressing an urge to act. Traumatic brain injury (TBI) can significantly impair the brain's ability to voluntarily stop or inhibit certain actions. Using brain imaging (functional magnetic resonance imaging, or fMRI) and brain stimulation (transcranial magnetic stimulation, or TMS) to investigate how people perform activities that involve moving and suppressing movements, researchers hope to better understand how these brain areas might be affected in people who have had TBI.

Objectives:

* To determine the parts of the brain involved in suppressing an urge to act.
* To determine the extent to which traumatic brain injury affecting certain parts of the brain is involved in problems with suppressing an urge to move and stopping movement.

Eligibility:

- Individuals 18 to 40 years of age who have had mild or moderate TBI, or are healthy volunteers.

Design:

* This research study includes a screening visit and two study visits, each of which will last at least 2 hours.
* Participants will be screened with a physical examination and medical history. Women who can become pregnant will have a urine pregnancy test before being allowed to participate in the study.
* At the first study visit, participants will complete one of the following experiment tests in an MRI scanner.
* Experiment 1: Participants will be shown arrows or images on a computer screen, and will press a button or not press a button depending on the image shown. Participants will practice the experiment tasks before performing them during MRI scans.
* Experiment 2: Participants will be shown arrows or images on a computer screen, and will press a button or not press a button depending on the image shown. Participants will also have TMS while at rest, and will perform the experiment tasks during the MRI scan.
* At the second study visit, participants will have an fMRI scan where they will be asked to do simple response tasks with a computer outside the MRI scanner.

Background:

- Previous research has shown that certain parts of the brain are involved in voluntarily stopping an ongoing motor response (movement); however, it is not known whether this same network is also involved in suppressing an urge to act. Traumatic brain injury (TBI) can significantly impair the brain's ability to voluntarily stop or inhibit certain actions. Using brain imaging (functional magnetic resonance imaging, or fMRI) and brain stimulation (transcranial magnetic stimulation, or TMS) to investigate how people perform activities that involve moving and suppressing movements, researchers hope to better understand how these brain areas might be affected in people who have had TBI.

Objectives:

* To determine the parts of the brain involved in suppressing an urge to act.
* To determine the extent to which traumatic brain injury affecting certain parts of the brain is involved in problems with suppressing an urge to move and stopping movement.

Eligibility:

- Individuals 18 to 40 years of age who have had mild or moderate TBI, or are healthy volunteers.

Design:

* This research study includes a screening visit and two study visits, each of which will last at least 2 hours.
* Participants will be screened with a physical examination and medical history. Women who can become pregnant will have a urine pregnancy test before being allowed to participate in the study.
* At the first study visit, participants will complete one of the following experiment tests in an MRI scanner.
* Experiment 1: Participants will be shown arrows or images on a computer screen, and will press a button or not press a button depending on the image shown. Participants will practice the experiment tasks before performing them during MRI scans.
* Experiment 2: Participants will be shown arrows or images on a computer screen, and will press a button or not press a button depending on the image shown. Participants will also have TMS while at rest, and will perform the experiment tasks during the MRI scan.
* At the second study visit, participants will have an fMRI scan where they will be asked to do simple response tasks with a computer outside the MRI scanner.

DETAILED DESCRIPTION:
Objectives

Voluntarily stopping an on-going motor response has been shown to engage a specific prefrontal-basal-ganglia (PBG) neural network. However, it is not known whether the PBG network is also crucial for other types of response inhibition such as suppressing an urge to act (i.e., habitual impulse), a common impairment after traumatic brain injury (TBI). The objectives of this protocol are: 1) to determine whether the PBG network is engaged in suppressing habitual impulses and, 2) to determine the extent to which the (PBG) neural network can account for the deficiency in response inhibition after mild to moderate traumatic brain injury (TBI). The proposed studies will involve performance of simple behavioral tasks, functional magnetic resonance imaging (fMRI), transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), and diffusion tensor imaging (DTI). tDCS will be applied separately from fMRI scans. TMS will be applied separately or concurrently during fMRI scans.

Study Population

One hundred and ninety healthy adult volunteers and 95 patients with mild to moderate TBI will be recruited under the protocol. Eighty of the healthy volunteers and 80 of the patients will be recruited under the project funded by the Center for Neuroscience and Rehabilitative Medicine (CNRM) at the Uniformed Services University of the Health Sciences (USUHS).

Design

There are five experiments. Experiment 1 includes healthy adult volunteers and mild to moderate TBI patients to determine whether the PBG inhibitory network is engaged in the suppression of an undesirable habitual impulse. Subjects will perform simple motor response tasks during fMRI scans. Experiment 2 will use fMRI with behavioral tasks and apply single-pulse TMS during fMRI scans when subjects are at rest to examine whether changes in the active and resting neural connectivity within the PBG network are associated with deficiency in response inhibition after mild to moderate TBI. Experiment 3 will involve only healthy volunteers to determine the effect of disruption of critical links/brain regions within the PBG network on response inhibition. Inhibitory rTMS (i.e., 1Hz repetitive TMS with stimulation intensity at 80% of a subject s own resting motor threshold [rMT]) will be applied in separate groups of subjects immediately before the behavioral tasks. Experiments 4-5 will use similar response tasks as in Experiment 1 but with patients who have had blast induced concussion(s). tDCS will be applied in Experiment 5 to examine the extent to which tDCS may change connectivity and improve rapid response inhibition. Additional behavioral measures, DTI, and high-resolution structural MRI images will be acquired in a separate session for all subjects.

Outcome Measures

Major outcome measures will include: 1) Task and TMS induced fMRI BOLD signal change and, 2) Behavioral performance data (reaction time and accuracy). Secondary measures: White matter fiber integrity and fiber tracking based on diffusion tensor imaging data.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 to 40
  2. Able to give consent
  3. Normal clinical examination for healthy subjects
  4. Must be able to follow instructions and perform required tasks, and TBI patients must have the Mini-mental state examination (MMSE) score of 25 or above.
  5. Clearly right dominant handedness as assessed by Handedness scales

MILD TBI:

Traumatically induced physiological disruption of brain function, as manifested by at least on the following:

1. Any loss of consciousness
2. Any loss of memory for events immediately before or after the accident (except for short-lasting benzodiazepines for sleep.
3. Focal neurological deficit(s) that may or may not be transient
4. Any alteration in metal state at the time of the accident (e.g. feeling dazed, disoriented or confused) and focal neurological deficit (s) that may or may not be transient, but where the severity of the injury does not exceed the following:

   * Loss of consciousness (LOC) of approximately 30 min
   * After 30 min, an initial Glasgow Coma Scale (GCS) sore of 13 - 15 (or clinically diagnosed concussion) and
   * Post-traumatic amnesia (PTA) not greater than 24 hour

Moderate TBI:

Those meeting the same criteria as mild TBI plus any one of the following:

1. GCS of 9-12 (if available) or results of a clinical evaluation as moderate TBI
2. Mental status change or LOC 30 min to 24 hour
3. PTA 1-7 days

EXCLUSION CRITERIA:

1. Being diagnosed as an alcoholic or with drug addiction.
2. Chronic use of medications acting primarily on the central nervous system such as those for seizures (e.g., carbamazepine, phenytoin) except for short-lasting benzodiazepines for sleep and antidepressants (e.g., SSRIs and SNRIs).
3. Pregnancy
4. Medical or technical contraindications to MRI procedures or devices producing artifacts that impair MRI signal (e.g., dental braces, pacemakers, implanted medication pumps, cochlear devices, neural stimulators, certain metals in the cranium, surgical clips, and other metal/magnetic implants, claustrophobia)
5. History of epilepsy (to avoid brain abnormalities other than mild to moderate TBI)
6. Less than three months post-TBI and with severe post traumatic stress disorder (PTSD) or PTSD Check List (PCL) score > 60
7. Penetrating head wound
8. For healthy volunteer, history of brain injury and/or structural MRI abnormality.
9. Staff from our section

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2010-08-10; Study Completion 2017-11-16

PRIMARY OUTCOMES:
Task-dependent and independent fMRI BOLD signal | Ongoing
TMS effects on behavioral performance | Ongoing

SECONDARY OUTCOMES:
Behavioral performance data (reaction time and accuracy) | Ongoing
White matter fiber integrity in TBI patients estimated by the degree of fractional anisotropy (FA) from diffusion tensor imaging (DTI) signals. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson JR. Automaticity and the ACT* theory. Am J Psychol. 1992 Summer;105(2):165-80. PMID 1621879
- [Background] Aron AR, Poldrack RA. Cortical and subcortical contributions to Stop signal response inhibition: role of the subthalamic nucleus. J Neurosci. 2006 Mar 1;26(9):2424-33. doi: 10.1523/JNEUROSCI.4682-05.2006. PMID 16510720
- [Background] Aron AR, Behrens TE, Smith S, Frank MJ, Poldrack RA. Triangulating a cognitive control network using diffusion-weighted magnetic resonance imaging (MRI) and functional MRI. J Neurosci. 2007 Apr 4;27(14):3743-52. doi: 10.1523/JNEUROSCI.0519-07.2007. PMID 17409238